CLINICAL TRIAL: NCT03322787
Title: Effect of Exercise Training Under High Flow Oxygen (HFO) Device on Endurance Tolerance in Patients With COPD and Chronic Respiratory Failure: a Randomized Controlled Study.
Brief Title: Effect of Exercise Training Under HFO Device on Endurance Tolerance in Patients With COPD and CRF: a Randomized Controlled Study.
Acronym: HFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Azienda Ospedaliera Ospedale Maggiore di Crema (Other); University of Modena and Reggio Emilia (Other); Villa Pineta Hospital (Other); Fisher and Paykel Healthcare (Industry); Associazione Riabilitatori Insufficienza Respiratoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: ICS Maugeri - CE2109
Record Dates: First submitted 2017-10-03; First posted 2017-10-26 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oxygen (No Intervention): The training will be performed using oxygen by the Venturi mask with the FiO2 set during the run - in session.
- HFO (Experimental): The training will be performed using the HFO device during the run - in session at iso_FiO2 as in the Control Group (Oxygen by Venturi mask).
  Interventions: Device: HFO

INTERVENTIONS:
Device: HFO — Training will be done using the HFO device. Air-flow will set at the highest value tolerated by the patients, until a maximum value of 60 l/min permitted and FiO2 set during the run-in. The HFO will be administered using the AIRVO2® (Fisher&Paykel- NewZealand). Afterwards, the oxygen flow provided into the system will be progressively increased until the pre-fixed FiO2 will be reached, as displayed by the AIRVO2 monitor.
  Arms: HFO

SUMMARY:
Current literature clearly shows the benefit of pulmonary rehabilitation in symptomatic COPD (Trooster,2005). However, these patients are frequently unable to sustain a work-load sufficiently high to obtain a full benefit on exercise tolerance (Trooster,2005). Especially in patients with Chronic Respiratory Failure (CRF), the development of hypoxia (O'Donnel,2001) and the increase of dead space (Elbehairy,2015) during effort explain the out-of-proportion increase in ventilation leading to an early achievement of the ventilatory reserve. Recent studies on heated and humidified high flow oxygen (HFO) delivered through nasal cannula, show several positive effects on breathing pattern and ventilatory efficiency, mostly in critical care setting and at rest (Spoletini,2015). Some recent physiological studies have evidenced that high flows of humidified oxygen improve exercise performance in patients with COPD and severe oxygen dependency, in part by enhancing oxygenation (Chatila,2004). Recently, a pilot study by our group showed that HFO may improve the exercise performance in severe COPD patients with ventilatory limitation. This effect is associated to an improvement of oxygen saturation (SatO2) and perceived symptoms at iso-time (Cirio,2016). No clinical studies are available about the use of HFO during exercise training. The investigators hypothesize that, in severe COPD patients with CRF and exercise limitation , the use of HFO could improve the efficiency of ventilation, leading to an increase in the patient's exercise performance and outcome.

Primary aim will be to evaluate in patients COPD with CRF the difference in the endurance tolerance improvement (expressed in minutes) after an high intensity training program, at iso-FiO2, using HFO with respect to usual oxygen administration by " Venturi Mask" .

Secondary objectives will be to study effectiveness of HFO with respect to "Venturi Mask" in terms of improvement of meters of 6 Minute Walking Test, dyspnea at rest, peripheral and respiratory muscle strength,blood gases, motor and respiratory disability,quality of life,impact of the disease and patients satisfaction.

DETAILED DESCRIPTION:
160 patients will be enrolled in 4 different hospitals. One of those, ICS Maugeri, will contribute with 5 different Institutes [Brescia, Pavia, Tradate (VA),Veruno (NO) and Cassano delle Murge (BA)]. Thus the total recruiting centers will be eight.

During the whole rehabilitation period, the patients will perform one training session/day.

The patients will use medications and oxygen therapy at rest as prescribed. The patients will perform no less than 20 training sessions within a period of one month. The rehabilitative intervention will be constantly supervised by a respiratory therapist.

The cycle load started from the 50% of the theoretical maximum watt (evaluated by 6 minutes walking test [6MWT] through the Luxton's equation) (Luxton,2008) and increased by Maltais's protocol (Maltais,1997). Run-in training session: all patients will be submitted to a preliminary 30 minute training under a Venturi mask to set the FiO2 able to maintain SpO2 constantly up to 93%. Usual nocturnal ventilation and nocturnal oxygen therapy under nasal cannula will be allowed.

Patients will be randomized to 2 groups:

* OXYGEN (Control Group, n = 80): the training will be performed using the Venturi mask with the FiO2 set during the run -in session.
* HFO (TREATMENT Group, n = 80): the training will be performed using the HFO device. Air-flow will be set at the highest value tolerated by the patient, until a maximum value of 60 l/min and with the same FiO2 set of the Control Group (iso-FiO2) during the run-in session.

The HFO will be administered using the AIRVO2® (Fisher&Paykel- NewZealand, CE0123 - 93/42/CEE). Afterwards, the oxygen flow provided into the system will be progressively increased until the pre-fixed FiO2 will be reached, as displayed by the AIRVO2 monitor.

the investigators will expect an enrollmnet rate of at least 23 patients/center. An enrollment rate less than 12 patients/center will not guarantee 1 author name on the possible Scientific publication. All the centers will be named in a possible congress/poster presentation. The possible publication will consider that a) the study is under the endorsement of AIPO and ARIR societies and b) Authors acknowledge the Industry contribution.

Measures

At baseline (T0), for both groups the following clinical evaluations will be performed:

* Anthropometric (age, BMI, diagnosis)
* Scale of comorbidity (CIRS)
* Spirometry (FEV1 %prd, FVC %prd, FEV1/FVC)

At baseline (T0) and at the end of rehabilitative program (T1), an operator, unblinded to the study, will perform the following outcome measures:

* Constant load cycle-ergometer endurance [at work load of 80% of maximal load predicted by Luxon's equation (Luxton,2008)] under usual oxygen supply with nasal cannula
* Arterial blood gas analysis (ABG) under room air
* 6-min walking test (6MWT) under usual oxygen supply with nasal cannula
* Scale of the MRC dyspnea
* Quality of Life (MRF26 scale)
* Respiratory muscle strength (MIP and MEP)
* Biceps and Quadriceps muscle strength tested by manual dynamometer and MRC muscle scale
* Disability (Barthel index, Barthel dispnea)
* Impact of the disease (CAT scale)

During each training session the investigators will evaluate:

* Side effects (discomfort, severe dyspnea, dryness of mucosa , etc)
* delta increase in training prescription (% of variation in watts compared with the previous session)

Only at the end of the program (T1) the investigators will evaluate :

1. patient satisfaction for training sessions with a Likert scale (0= no discomfort; 1 minimum discomfort; 2= moderate discomfort; 3 = high discomfort; 4= maximum discomfort)
2. drops out (number and reasons: exacerbation, intolerance of treatment, refuse, early discharge, etc)

Statistical analysis will be performed using STATA 12. Descriptive data will be shown as mean ± SD.

The analyses will be conducted on a intention-to-treat (all randomized patients) or per-protocol (all completers) basis. A two-sample t test was used to explore differences in: 1. baseline characteristics intervention and control groups, 2. between improvers and non improvers, 3.between completers and 4. dropouts and to assess differences in changes of parameters following the rehabilitation program between intervention and control groups. Wilcoxon matched-paired tests and Mann-Whitney U test will be employed for nonparametric data. Frequency distributions will be analyzed with χ2 test. Data will be considered significant for p<0.05.

The sample estimated size for two sample comparison of means on primary outcome (endurance time evaluated by cicloergometer at costant load) (alpha error 0.05, beta error=0.90 considering mean control group=150 s, mean treatment group=280s, standard deviation for both groups 250s ) is 156 patients

ELIGIBILITY:
Inclusion Criteria:

* COPD and CRF diagnosis under LTOT,
* clinical stability (pH > 7.35 and < 7.46, no change in respiratory drugs therapy during the last seven days)

Exclusion Criteria:

* orthopedic or neurological disease,
* cognitive impairment (Mini Mental State Examination < 22)
* anamnestic history of ischemic heart disease or heart failure, COPD+ fibrosis and COPD+ OSAS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness on endurance tolerance | At Baseline
  To evaluate the difference in the endurance tolerance improvement (endurance time) with a costant load cycloergometer test.

SECONDARY OUTCOMES:
Effectiveness on functional capacity | At 1 month
  To evaluate effectiveness of HFO with respect to "Venturi Mask" in terms of improvement of meters at 6-min walking test.
Effectiveness on dyspnea | At 1 month
  To evaluate effectiveness of HFO with respect to "Venturi Mask" in terms of dyspnea evaluation, MRC scale for dyspnea will be used.
Effectiveness on respitarory muscle strength | At 1 month
  To evaluate effectiveness of HFO with respect to "Venturi Mask" in terms of improvement in respiratory muscle strenght measured by MIP/MEP.
Effectiveness on peripheral muscle strenght | At 1 month
  To evaluate effectiveness of HFO with respect to "Venturi Mask" in terms of improvement in peripheral muscles [biceps and quadriceps] evaluated by manual dinamometer and MRC muscle scale.
Effectiveness on blood gases | At one month
  To evaluate improvement of blood gases (PaO2/FiO2 PaCO2, pH) arterial blood gases analysis will be used.
Effectiveness on disability | At 1 month
  To evaluate disability of HFO with respect to "Venturi Mask" , disability will be measured by Barthel index and Barthel Dyspnea.
Effectiveness on quality of life | At 1 month
  To evaluate quality of life MRF-26 will be used.
Effectiveness on impact of the disease | At 1 month
  To evaluate impact of disease CAT will be used.
Effectivenes on satisfaction | At 1 month
  Patient satisfaction for training session will be assessed by a Likert scale 0-4 (0= no discomfort; 1= minimum discomfort; 2=moderate discomfort; 3= high discomfort; 4= maximum discomfort).

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vitacca, MD, Principal Investigator — ICS Maugeri Lumezzane
Locations (1):
- ICS Maugeri, IRCCS Lumezzane, Lumezzane, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Troosters T, Casaburi R, Gosselink R, Decramer M. Pulmonary rehabilitation in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 Jul 1;172(1):19-38. doi: 10.1164/rccm.200408-1109SO. Epub 2005 Mar 18. No abstract available. PMID 15778487
- [Background] O'Donnell DE, D'Arsigny C, Webb KA. Effects of hyperoxia on ventilatory limitation during exercise in advanced chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Mar;163(4):892-8. doi: 10.1164/ajrccm.163.4.2007026. PMID 11282762
- [Background] Elbehairy AF, Ciavaglia CE, Webb KA, Guenette JA, Jensen D, Mourad SM, Neder JA, O'Donnell DE; Canadian Respiratory Research Network. Pulmonary Gas Exchange Abnormalities in Mild Chronic Obstructive Pulmonary Disease. Implications for Dyspnea and Exercise Intolerance. Am J Respir Crit Care Med. 2015 Jun 15;191(12):1384-94. doi: 10.1164/rccm.201501-0157OC. PMID 25826478
- [Background] Spoletini G, Alotaibi M, Blasi F, Hill NS. Heated Humidified High-Flow Nasal Oxygen in Adults: Mechanisms of Action and Clinical Implications. Chest. 2015 Jul;148(1):253-261. doi: 10.1378/chest.14-2871. PMID 25742321
- [Background] Chatila W, Nugent T, Vance G, Gaughan J, Criner GJ. The effects of high-flow vs low-flow oxygen on exercise in advanced obstructive airways disease. Chest. 2004 Oct;126(4):1108-15. doi: 10.1378/chest.126.4.1108. PMID 15486371
- [Background] Cirio S, Piran M, Vitacca M, Piaggi G, Ceriana P, Prazzoli M, Paneroni M, Carlucci A. Effects of heated and humidified high flow gases during high-intensity constant-load exercise on severe COPD patients with ventilatory limitation. Respir Med. 2016 Sep;118:128-132. doi: 10.1016/j.rmed.2016.08.004. Epub 2016 Aug 8. PMID 27578482
- [Background] Luxton N, Alison JA, Wu J, Mackey MG. Relationship between field walking tests and incremental cycle ergometry in COPD. Respirology. 2008 Nov;13(6):856-62. doi: 10.1111/j.1440-1843.2008.01355.x. PMID 18811884
- [Background] Maltais F, LeBlanc P, Jobin J, Berube C, Bruneau J, Carrier L, Breton MJ, Falardeau G, Belleau R. Intensity of training and physiologic adaptation in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1997 Feb;155(2):555-61. doi: 10.1164/ajrccm.155.2.9032194.
- [Background] Shah S, Vanclay F, Cooper B. Improving the sensitivity of the Barthel Index for stroke rehabilitation. J Clin Epidemiol. 1989;42(8):703-9. doi: 10.1016/0895-4356(89)90065-6. PMID 2760661
- [Background] Vitacca M, Paneroni M, Baiardi P, De Carolis V, Zampogna E, Belli S, Carone M, Spanevello A, Balbi B, Bertolotti G. Development of a Barthel Index based on dyspnea for patients with respiratory diseases. Int J Chron Obstruct Pulmon Dis. 2016 Jun 7;11:1199-206. doi: 10.2147/COPD.S104376. eCollection 2016. PMID 27354778
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Vidotto G, Carone M, Jones PW, Salini S, Bertolotti G; Quess Group. Maugeri Respiratory Failure questionnaire reduced form: a method for improving the questionnaire using the Rasch model. Disabil Rehabil. 2007 Jul 15;29(13):991-8. doi: 10.1080/09638280600926678. PMID 17612984
- [Background] Linn BS, Linn MW, Gurel L. Cumulative illness rating scale. J Am Geriatr Soc. 1968 May;16(5):622-6. doi: 10.1111/j.1532-5415.1968.tb02103.x. No abstract available. PMID 5646906
- [Derived] Vitacca M, Paneroni M, Zampogna E, Visca D, Carlucci A, Cirio S, Banfi P, Pappacoda G, Trianni L, Brogneri A, Belli S, Paracchini E, Aliani M, Spinelli V, Gigliotti F, Lanini B, Lazzeri M, Clini EM, Malovini A, Ambrosino N; Associazione Italiana Riabilitatori Insufficienza Respiratoria and Associazione Italiana Pneumologi Ospedalieri rehabilitation group. High-Flow Oxygen Therapy During Exercise Training in Patients With Chronic Obstructive Pulmonary Disease and Chronic Hypoxemia: A Multicenter Randomized Controlled Trial. Phys Ther. 2020 Aug 12;100(8):1249-1259. doi: 10.1093/ptj/pzaa076. PMID 32329780